CLINICAL TRIAL: NCT07057804
Title: Role of Lung and Diaphragm Ultrasound in Predicting Extubation and Weaning of Mechanically Ventilated Patients in Intensive Care Unit
Brief Title: Lung and Diaphragm Ultrasound in Predicting Extubation and Weaning of Mechanically Ventilated Patients in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Mabrouk Elsayed Ibrahim, Resident at Anesthesia, Surgical Intensive Care and Pain Management, Faculty of Medicine, Kafr Elsheikh University, Kafr Elsheikh, Egypt., Kafrelsheikh University
Other Study IDs: KFSIRB200-202
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Lung; Diaphragm; Ultrasound; Extubation; Weaning; Mechanically Ventilation; Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients who met the standard clinical weaning criteria underwent bedside lung and diaphragm ultrasound at the end of a successful spontaneous breathing trial (SBT).
  Interventions: Diagnostic Test: Lung Ultrasound; Diagnostic Test: Diaphragm Ultrasound

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound — Ultrasound was performed at the bedside with the patient in a semi-recumbent position using a 3.5-5 MHz curvilinear probe. Lung ultrasound was conducted across 12 zones (anterior and posterior) to evaluate aeration and calculate the lung ultrasound score (LUS).
Diagnostic Test: Diaphragm Ultrasound — Ultrasound was performed at the bedside with the patient in a semi-recumbent position using a 3.5-5 MHz curvilinear probe. Diaphragmatic excursion and thickening fraction were measured on the right hemidiaphragm.

SUMMARY:
This study aims to evaluate the role of lung ultrasound score (LUS), diaphragmatic excursion (DE), and diaphragmatic thickening fraction (DTF) as predictors of successful extubation in mechanically ventilated patients in the intensive care unit (ICU). It also compares these ultrasound-based parameters to traditional weaning criteria.

DETAILED DESCRIPTION:
Mechanical ventilation is a necessary life support technology for critically ill patients. The weaning outcome affects the morbidity and mortality of patients when their primary disease improves.

Moreover, lung ultrasonography can be used as an effective measure in the evaluation of lung aeration which is useful during the weaning procedure as it reflect the aeration loss and consequently predict the respiratory distress in the postintubation period, a validated score termed the lung ultrasound score(LUS) can be used to evaluate the loss of lung aeration.

Numerous data measured through diaphragmatic ultrasonography have been recommended for the same purpose, which involve measurement of diaphragmatic muscle movement during inspiration or excursion during the respiratory cycle (DE), and diaphragmatic muscle thickening or diaphragmatic thickening fraction (DTF).

ELIGIBILITY:
Inclusion Criteria:

* All patients who will meet the following weaning criteria undergo Spontaneous Breathing Trial, which include,

  * Improvement of disease acute phase which necessitated mechanical ventilation.
  * Stable neurological status.
  * No hemodynamic instability (heart rate ≤ 120/min, systolic blood pressure higher than 90 mmHg and lower than 160 mmHg) in the absence of any vasoactive support therapy.
  * PaO2>60 mm Hg or SaO2 ≥ 90% or more with FiO2 ≤ 0.4.
  * Afebrile and there were no significant abnormalities in the electrolyte levels.

Exclusion Criteria:

* Hemodynamic unstable patients
* Patients with severe intracranial disease,
* Tracheostomy.
* Severe intensive care unit (ICU) acquired neuromyopathy, with primary unilateral/bilateral absence of diaphragmatic mobility,
* Patients who had previously failed spontaneous breathing trial (SBT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study trial was carried out on 90 patients required invasive mechanical ventilation for a minimum of 24 hours and weaning criteria.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Success rate of extubation | 48 hours post-extubation
  Success rate of extubation was recorded

SECONDARY OUTCOMES:
Diaphragmatic Excursion (DE) | Within 1 hour prior to extubation
  Assessment of diaphragmatic excursion as a predictor of weaning success, measured using ultrasound.
Diaphragmatic Thickening Fraction (DTF) | Within 1 hour prior to extubation
  Assessment of diaphragmatic Thickening Fraction (DTF) as a predictor of weaning success, measured using ultrasound.
Lung Ultrasound Score (LUS) | Within 1 hour prior to extubation
  Evaluation of lung Ultrasound Score (LUS) as a predictor of extubation outcome, measured before extubation using standard lung ultrasound protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr Elsheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.